CLINICAL TRIAL: NCT00005253
Title: Proarrhythmic Medicines and Primary Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1135; R01HL042456 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2006-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Heart Arrest; Hypertension; Arrhythmia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Arrest; Hypertension; Arrhythmias, Cardiac

SUMMARY:
To determine whether treatment with antidepressant, anticonvulsant, and antiarrhythmic drug therapies having the potential for proarrhythmia increased the risk of primary cardiac arrest. The aim of the original grant, starting in 1990 and ending in 1994, was to determine whether use of diuretics for hypertension increased the risk of primary cardiac arrest compared to the use of other antihypertensive agents.

DETAILED DESCRIPTION:
BACKGROUND:

The original grant from 1990 to 1995 was funded because analyses of clinical trial subgroups had raised the concern that, in patients with high blood pressure, diuretic therapy may increase the risk of sudden cardiac death. Given the size of the hypertensive population in the United States, the prevalence of diuretic therapy for hypertension, and the persistent concerns regarding the relation of diuretic therapy to the risk of primary cardiac arrest (PCA), the study proved to be of particular interest to clinicians, epidemiologists, public policy makers, and the general public.

Beginning in 1995 when the grant was renewed, unexpected findings from the Cardiac Arrhythmia Suppression Trial--an adverse effect on mortality of two antiarrhythmic drug therapies--had heightened concerns that drug therapies other than diuretics may increase the risk of primary cardiac arrest.

DESIGN NARRATIVE:

The original study beginning in 1990 was population-based with a case-control design. Using the community-based surveillance system for out-of-hospital primary cardiac arrest in Seattle and King County, Washington, all cases of primary cardiac arrest (PCA) were identified which had occurred among 18,000 pharmacologically-treated hypertensive patients receiving care at Group Health Cooperative (GHC) from 1977-1993. Approximately 180 cases were identified. Controls were obtained from a random sample of GHC enrollees with pharmacologically-treated hypertension, matched to cases at a ratio of 3 to 1, according to age, gender, and year of occurrence of PCA. The computerized pharmacy data base of GHC allowed ascertainment of patterns of exposure to specific antihypertensive drug therapy in an identical fashion for both cases and controls. Medical records were reviewed to gather information about potential confounding factors and effect modifiers, such as severity of hypertension. Data analysis, using stratification and logistic regression, determined whether use of diuretics increased the risk of PCA compared to use of other antihypertensive agents; whether the risk of PCA depended upon the dose of diuretic therapy; and whether electrocardiographic abnormalities modified the risk of PCA associated with diuretics.

The study was renewed in 1995 to determine whether treatment with antidepressant, anticonvulsant, and antiarrhythmic drug therapies having the potential for proarrhythmia increased the risk of primary cardiac arrest. The study was a population-based case-control study nested within a cohort of patients who received medical care at a large pre-paid Health Care Plan in Seattle, Washington. Cases were patients who had a primary cardiac arrest between 1977 to 1994. Controls were a stratified random sample of patients, frequency-matched to cases by age, gender, calendar-year, and known heart disease. Treatment with drugs was assessed through a computerized pharmacy database. Ambulatory-care medical records were reviewed to assess clinical characteristics, including the indication for therapy, the severity of heart disease, co-existing morbidity, and other risk factors. For both antidepressant and anticonvulsant drugs, analyses were stratified by known heart disease, because the risk of treatment might be particularly large among patients with known heart disease. For antiarrhythmic drugs, analyses were restricted by a single, current indication for the therapy--maintenance of sinus rhythm among patients with chronic atrial fibrillation; and, by the availability of a prior echocardiogram, in order to control for the type and severity of underlying heart disease. After adjustment for potential confounders, the investigators estimated the relative safety of: 1) drugs within the same therapeutic class; and, 2) the dosage schedule for specific drugs. In addition, they determined if concurrent treatment with other drugs that altered cardiac conduction or morbidity that altered drug disposition influenced the risk among patients treated with a drug therapy.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-01; Study Completion 2000-01

CONTACTS AND LOCATIONS:
Overall Officials: David Siscovick — University of Washington

REFERENCES:
- [Background] Siscovick DS, Raghunathan TE, Psaty BM, Koepsell TD, Wicklund KG, Lin X, Cobb L, Rautaharju PM, Copass MK, Wagner EH. Diuretic therapy for hypertension and the risk of primary cardiac arrest. N Engl J Med. 1994 Jun 30;330(26):1852-7. doi: 10.1056/NEJM199406303302603. PMID 8196728
- [Background] Siscovick DS, Raghunathan TE, Rautaharju P, Psaty BM, Cobb LA, Wagner EH. Clinically silent electrocardiographic abnormalities and risk of primary cardiac arrest among hypertensive patients. Circulation. 1996 Sep 15;94(6):1329-33. doi: 10.1161/01.cir.94.6.1329. PMID 8822988
- [Background] Siscovick DS, Raghunathan TE, Psaty BM, Koepsell TD, Cobb L, Rautaharju PM, Wagner EH. Diastolic blood pressure and the risk of primary cardiac arrest among pharmacologically treated hypertensive patients. J Gen Intern Med. 1996 Jun;11(6):350-6. doi: 10.1007/BF02600046. PMID 8803741
- [Background] Rea TD, Siscovick DS, Psaty BM, Pearce RM, Raghunathan TE, Whitsel EA, Cobb LA, Weinmann S, Anderson GD, Arbogast P, Lin D. Digoxin therapy and the risk of primary cardiac arrest in patients with congestive heart failure: effect of mild-moderate renal impairment. J Clin Epidemiol. 2003 Jul;56(7):646-50. doi: 10.1016/s0895-4356(03)00075-1. PMID 12921933
- [Background] Empana JP, Jouven X, Lemaitre RN, Sotoodehnia N, Rea T, Raghunathan TE, Simon G, Siscovick DS. Clinical depression and risk of out-of-hospital cardiac arrest. Arch Intern Med. 2006 Jan 23;166(2):195-200. doi: 10.1001/archinte.166.2.195. PMID 16432088